CLINICAL TRIAL: NCT01529112
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of Oral E7080 in Addition to Best Supportive Care (BSC) Versus BSC Alone in Patients With Locally Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer Who Have Failed at Least Two Systemic Anticancer Regimens
Brief Title: A Study Comparing the Combination of the Best Supportive Care Plus E7080 Versus Best Supportive Care Alone, in Patients With Advanced Lung Cancer or Lung Cancer That Has Spread, Who Have Been Previously Treated, Unsuccessfully, With at Least 2 Different Treatments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E7080-703
Record Dates: First submitted 2012-01-06; First posted 2012-02-08 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Locally Advanced; Metastatic Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — lenvatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenvatinib (Experimental): Participants received lenvatinib 24 mg orally, once daily continuously in each 28-day treatment cycle plus Best Supportive Care (BSC)
  Interventions: Drug: Lenvatinib; Drug: BSC
- Lenvatinib matched placebo (Placebo Comparator): Participants received lenvatinib matched placebo orally, once daily continuously in each 28-day treatment cycle plus BSC
  Interventions: Drug: Lenvatinib matched placebo; Drug: BSC

INTERVENTIONS:
Drug: Lenvatinib
  Other Names: E7080
  Arms: Lenvatinib
Drug: Lenvatinib matched placebo
  Arms: Lenvatinib matched placebo
Drug: BSC

SUMMARY:
The purpose of this study is to compare the overall survival of patients receiving E7080 + Best Supportive Care (BSC) with those receiving placebo + Best Supportive Care.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled, multicenter, randomized Phase II study will consist of a 2-arm design, comparing E7080 + BSC (Arm 1) with placebo + BSC (Arm 2). Participants will be randomized in the ratio of 2:1 to receive either E7080 or placebo in a blinded manner.

ELIGIBILITY:
Inclusion Criteria

1. Age greater than or equal to 18 years;
2. Participants with histologically or cytologically confirmed non-squamous NSCLC with locally advanced or metastatic disease based on Tumor, Node, Metastasis (TNM) staging according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual, Seventh Edition, who had failed at least two lines of systemic anticancer therapy for advanced or metastatic NSCLC (did not include adjuvant chemotherapy). In countries where erlotinib was approved and marketed for the treatment of NSCLC, participants must have received erlotinib treatment (or gefitinib for participants outside of the US) for their NSCLC if they had known EGFR-activating mutations. Participants of unknown EGFR status who had not received prior erlotinib (or gefitinib) should have been tested for EGFR-activating mutations prior to study entry. In countries where crizotinib was approved and marketed, participants must have received crizotinib treatment for NSCLC that was ALK-positive. Participants with ALK positive NCSLC or participants with KRAS mutations were not required to have prior treatment with erlotinib or gefitinib
3. Participants must have at least 1 site of measurable disease by the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v.1.1);
4. ECOG PS of 0 to 2;
5. Participants must have adequate renal function as evidenced by serum creatinine less than or equal to 1.5 x upper limit of normal (ULN) or calculated creatinine clearance greater than or equal to 30 mL/min per the Cockcroft and Gault formula;
6. Blood pressure must be well-controlled (less than or equal to140/90 mm Hg at Screening) with or without antihypertensive medication. Participants must have no history of hypertensive crisis or hypertensive encephalopathy;
7. Participants must have adequate bone marrow function as evidenced by absolute neutrophil count (ANC) greater than or equal to 1.5 x 109/L, hemoglobin greater than or equal to 9.0 g/dL, and platelet count greater than or equal to 100 x 109/L;
8. Participants must have adequate liver function as evidenced by bilirubin less than or equal to 1.5 times the ULN, and alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 x ULN (in the case of liver metastases, less than or equal to 5 x ULN).
9. Participants must have adequate coagulation system function as defined by prothrombin time/International normalized ratio (INR) less than or equal to 1.5 x ULN.
10. Male or female participants of child-producing potential must agree to use double barrier contraception, oral contraceptives, or avoidance of pregnancy measures during the study and for 90 days after the last day of treatment;
11. Females of childbearing potential must have a negative serum pregnancy test;
12. Females may not be breastfeeding;
13. Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria

1. Prior therapy with E7080 or other small molecule vascular endothelial growth factor inhibitors;
2. Presence of brain metastases, unless the participant has received adequate treatment at least 4 weeks prior to randomization, and is stable, asymptomatic, and off steroids for at least 4 weeks prior to randomization;
3. Meningeal carcinomatosis;
4. Received chemotherapy, targeted therapy, radiotherapy, surgery, or immunotherapy within the 21 days prior to commencing study treatment or have not recovered from all treatment-related toxicities to Grade less than or equal to 2, except for alopecia;
5. Received treatment with another investigational agent within the 30 days prior to commencing study treatment or participants who have not recovered from side effects of an investigational drug to Grade less than or equal to 2, except for alopecia;
6. Participants with proteinuria greater than 1+ on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with 24-hour urine protein greater than or equal to 1 g/24 hours will be ineligible;
7. Serious non-healing wound, ulcer, bone fracture, or have undergone a major surgical procedure, open biopsy, or significant traumatic injury within the 28 days prior to commencing study treatment.
8. Major surgery scheduled during the projected course of the study;
9. History of bleeding diathesis or coagulopathy;
10. Active hemoptysis (defined as bright red blood of a half teaspoon or more) within the 30 days prior to study entry;
11. Refractory nausea and vomiting, malabsorption, significant bowel resection, or any other medical condition that would preclude adequate absorption or result in the inability to take oral medication;
12. Other malignancy within 3 years of randomization, with the exception of adequately treated carcinoma in situ of the cervix or non-melanoma skin cancer, with no subsequent evidence of recurrence and/or malignancies diagnosed at a stage where definitive therapy results in near certain cures.
13. Significant cardiovascular impairment (history of congestive heart failure New York Heart Association [NYHA] Class greater than II, unstable angina or myocardial infarction within the past 6 months, or serious cardiac arrhythmia);
14. Any history of cerebral vascular accident (CVA), transient ischemic attack (TIA), or Grade greater than or equal to 2 peripheral vascular disease unless they have had no evidence of active disease for at least 6 months prior to randomization;
15. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the 6 months prior to enrollment;
16. Participants with organ allografts requiring immunosuppression;
17. Known positive human immunodeficiency virus (HIV), known hepatitis B surface antigen, or hepatitis C positive;
18. Hypersensitivity to E7080 or any of the excipients;
19. Any history of or concomitant medical condition that, in the opinion of the Investigator, would compromise the participant's ability to safely complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2014-01-21 (Actual); Study Completion 2015-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harish Dave, Study Director — PharmaBio Development Inc.
Locations (50):
- United States (11):
  - Donald W. Hill, M.D., F.A.C.P., Casa Grande, Arizona
  - Arizona Oncology Associates , PC - HOPE, Tucson, Arizona
  - Ronald Yanagihara, MD 9360 North Name Uno Suite 130 Gilroy California 95020, Gilroy, California
  - Ocala Oncology Center, P.L., Ocala, Florida
  - Washington University 660 South Euclid Avenue Campus Box 8124 St Louis Missouri 63110, St Louis, Missouri
  - New York Oncology Heamatology - Latham, Clifton Park, New York
  - Montefiore Medical Park 1695 Easchester Road Floor 1 Bronx, NY 10461, New York, New York
  - Cancer Treatment and Research Centre Bismarck North Dakota 58501, Bismarck, North Dakota
  - Texas Oncology, P.A. - Paris, Paris, Texas
  - Texas Oncology, P.A. - Plano, Plano, Texas
  - Texas Oncology, P.A. - Waco, Waco, Texas
- Belgium (7):
  - OLV Ziekenhuis, Aalst
  - Grand Hopital de Charleroi, Charleroi
  - AZ Sint-Maarten, Duffel
  - UZ Antwerpen, Edegem
  - UZ Leuven, Leuven
  - C. H. R. de la Citadelle, Liège
  - Domaine Universitaire du Sart-Tilman, Liège
- Czechia (4):
  - Institut onkologie a rehabilitace Na Plesi, Nová Ves pod Pleší
  - Avicennus, s.r.o., Nymburk
  - Fakultni nemocnice Na Bulovce, Prague
  - Oblastni nemocnice Pribram, a.s., Příbram
- Hungary (7):
  - Semmelweis Egyetem AOK, Budapest
  - Orszagos Koranyi TBC es Pulmonologiai Intezet, Budapest
  - Matrai Gyogyintezet, Mátraháza
  - Fejer Megyei Szent Gyorgy Korhaz, Székesfehérvár
  - Komarom-Esztergom Megyei Onkorm. Szent Borbala Korhaza, Tatabánya
  - Tudogyogyintezet Torokbalint, Törökbálint
  - Zala Megyei Korhaz, Zalaegerszeg
- Italy (9):
  - Azienda Ospedaliera G. Rummo, Benevento
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Azienda Ospedaliera San Gerardo, Milan
  - Istituto Clinico Humanitas, Milan
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Fondazione Salvatore Maugeri IRCCS, Pavia
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Ospedale Mater Salutis, Verona
- South Korea (7):
  - Chungbuk National University Hospital, Chungcheongbuk-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea Yeouido St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- United Kingdom (5):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Southampton General Hospital, Southampton, Hampshire
  - North Staffs Royal Infirmary, Stoke-on-Trent, Staffordshire
  - Beatson West of Scotland Cancer Centre, Glasgow, Strathclyde
  - New Cross Hospital, Wolverhampton, West Midlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The participant flow is based on data cut-off date of 21 January 2014 as the study is ongoing.
Groups:
- Lenvatinib: Participants received lenvatinib 24 mg orally, once daily continuously in each 28-day treatment cycle.
- Lenvatinib Matched Placebo: Participants received lenvatinib matched placebo orally, once daily continuously in each 28-day treatment cycle.
Period: Overall Study
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Started | 89 | 46
Completed | 20 (On treatment=2, Discontinued treatment-continued follow-up=18 (data cut-off date 21 January 2014)) | 5 (Discontinued treatment-continued follow-up=5 (data cut-off date 21 January 2014))
Not Completed | 69 | 41
Not completed — Adverse Event | 2 | 0
Not completed — Death | 59 | 38
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo | Total
Number analyzed (Participants) | 89 | 46 | 135
Age, Continuous [Median (Full Range); unit: Years] | 63 [41 to 82] | 63.5 [44 to 77] | 63 [41 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 19 | 63
  Male | 45 | 27 | 72

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Treatment Emergent Non-serious Adverse Events (AEs) and Treatment Emergent Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered with an investigational product. A SAE was defined as any untoward medical occurrence that at any dose; resulted in death, was life-threatening (i.e., the subject was at a risk of death at the time of the event; this did not include an event that hypothetically might have caused death if it had been more severe), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, or was a congenital abnormality/birth defect. In this study, treatment emergent adverse events (TEAEs) (defined as an AE (serious/non-serious) that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication) were assessed.
Time Frame: For each participant, from the first dose till 30 days after the last dose or up to approximately 2 years (data cut-off date of 21 January 2014)
Population: Safety was analyzed in Safety Analysis Set defined as all subjects enrolled and randomized to treatment in study, except for those who (i) dropped out prior to receiving any study drug, or (ii) were without any safety assessment following the first dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 89 | 46
Participants
  Treatment Emergent Non-Serious AEs | 83 | 42
  Treatment Emergent SAEs | 46 | 21

2. Secondary Outcome: 6-Month Survival Rate
Description: Event-free survival rate was calculated using Kaplan Meier estimations. The percentage of participants with event free survival up to 6 months and the corresponding 95% confidence interval were estimated for each treatment group. The data presented is based on the data cut-off date of 26 November 2013 while the study is still ongoing.
Time Frame: From date of randomization (Day 1) up to 6 months
Population: The analysis was performed using the Intent-to-Treat Population, defined as all randomized subjects.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 89 | 46
Percentage of Participants | 61.6 [50.24 to 71.1] | 49 [33.49 to 62.8]

3. Secondary Outcome: 1-year Survival Rate
Description: Event-free survival rate was calculated using Kaplan Meier estimations. The percentage of participants with event free survival up to 1 year and the corresponding 95% confidence interval were estimated for each treatment group. The data presented is based on the data cut-off date of 26 November 2013 while the study is still ongoing.
Time Frame: From date of randomization (Day 1) up to 1 year
Population: The analysis was performed using the Intent-to-Treat Population, defined as all randomized subjects.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 89 | 46
Percentage of Participants | 35.8 [25.13 to 46.54] | 20.5 [9.96 to 33.74]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of the randomization until the date of first documented disease progression according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 or date of death from any cause (whichever occurred first), assessed based on investigator's assessment. Disease progression per RECIST v1.1 was defined as at least a 20% relative increase and 5 mm absolute increase in the sum of diameters of target lesions (taking as reference the smallest sum on study), recorded since the treatment started or the appearance of 1 or more new lesions. The data presented is based on the data cut-off date of 21 January 2014 while the study is still ongoing.
Time Frame: From date of randomization (Day 1) until date of first documentation of disease progression or death from any cause (whichever occurred first) or up to approximately 2 years (data cut-off date of 21 January 2014)
Population: The analysis was performed using the Intent-to-Treat Population, defined as all randomized subjects.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 89 | 46
weeks | 20.9 [15.86 to 23.86] | 7.9 [7.43 to 8.14]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR, defined as the percentage of participants who had best overall response (BOR) of complete response (CR) or partial response (PR) as determined by investigator using RECIST 1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. ORR = CR + PR. The data presented is based on the data cut-off date of 21 January 2014 while the study is still ongoing.
Time Frame: From date of randomization (Day 1) until disease progression or death, development of unacceptable toxicity, withdrawal of consent, withdrawal by Investigator, or up to approximately 2 years (data cut-off date of 21 January 2014)
Population: The analysis was performed using the Intent-to-Treat Population, defined as all randomized subjects.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 89 | 46
Percentage of Participants | 10.1 [4.7 to 18.3] | 2.2 [0.1 to 11.5]

6. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization until the date of death from any cause.
Time Frame: From date of randomization (Day 1) until occurrence of 90 deaths in the study (cut off date 26 November 2013), approximately 22 months
Population: The analysis was performed using the Intent-to-Treat Population, defined as all randomized subjects.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 89 | 46
weeks | 38.4 [26.57 to 47.86] | 24.1 [15.29 to 36.43]

7. Secondary Outcome: Response Duration (RD)
Description: Response duration, defined as the time from the date of the first assessment demonstrating a CR or PR to the date of the first assessment demonstrating progressive disease or death, whichever occurred first. This is an investigator assessed outcome, measured using RECIST 1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Response duration was summarized by including only subjects with events. The data presented is based on the data cut-off date of 21 January 2014 while the study is still ongoing.
Time Frame: as for outcome 5
Population: The analysis was performed using subjects with events.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 6 | 1
Weeks | 24.2 [12.71 to 33.14] | 43.3 [NA to NA] — Not applicable as there was only one participant with event.

8. Secondary Outcome: Disease Control Rate (DCR)
Description: The percentage of participants with CR, PR, or stable disease (SD) for greater than or equal to 12 weeks. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had to have reduction in short axis to less than 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable disease was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on the study. The data presented is based on the data cut-off date of 21 January 2014 while the study is still ongoing.
Time Frame: as for outcome 5
Population: The analysis was performed using the Intent-to-Treat Population, defined as all randomized subjects.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 89 | 46
Percentage of Participants | 42.7 [32.3 to 53.6] | 19.6 [9.4 to 33.9]

9. Secondary Outcome: The Percentage of Participants With The European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Symptom Scores Achieving Clinically Significant Deterioration on Quality of Life (QOL)
Description: The EORTC QLQ-C30 symptom score, a cancer specific self-reporting questionnaire was composed of 9-symptom scales assessing fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties. All of the multi-item scales and single-item measures ranged in score from 0 to 100. For each domain and item, a linear transformation was applied to standardize the raw score to a range from 0 to 100, with a higher scale score representing a higher response level/ high level of symptomatology / problems. The data is presented as percentage of participants with EORTC QLQ-C30 symptom score achieving clinically significant deterioration on QOL. Participants were considered as deteriorated for a given symptom if the change in score from Baseline was 10 points or higher at any time point after Baseline. The data presented is based on the data cut-off date of 21 January 2014 while the study is still ongoing.
Time Frame: Baseline (Day 1 of Cycle 1 (prior to treatment in Cycle 1)), every 4 weeks during treatment, and 4 weeks after completing treatment or up to approximately 2 years (data cut-off date of 21 January 2014)
Population: The analysis was performed using the Intent-to-Treat Population, defined as all randomized subjects.
Measure: Number; unit: Percentage of participants
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 89 | 46
Percentage of participants
  Appetite Loss (N=82, 39) | 59.8 | 66.7
  Constipation (N=82, 40) | 43.9 | 52.5
  Diarrhea (N=81, 40) | 48.1 | 17.5
  Dyspnea (N=82, 40) | 43.9 | 47.5
  Insomnia (N=82, 40) | 53.7 | 35
  Nausea and Vomiting (N=82, 40) | 46.3 | 40
  Pain (N= 82, 40) | 74.4 | 65
  Fatigue (N= 82, 40) | 63.4 | 67.5
  Financial Difficulties (N= 81, 40) | 34.6 | 30

10. Secondary Outcome: The Percentage of Participants With The European Organization for Research and Treatment of Cancer (EORTC) Module QLQ-LC13 (Lung Cancer 13) Symptom Scores Achieving Clinically Significant Deterioration on QOL
Description: The EORTC module QLQ-LC13 symptom score was a self-reporting cancer-specific questionnaire composed of 13 questions incorporated into 1 multi-item scale designed to evaluate dyspnea and a series of single items assessing different types of pain, as well as, cough, hemoptysis, dysphagia, sore mouth, alopecia, and peripheral neuropathy. For each domain and item, a linear transformation was applied to standardize the raw score to a range from 0 to 100, with 100 representing the best possible function/QOL, and highest burden of symptoms for symptom domains and single items. The data is presented as percentage of participants with EORTC module QLQ-C13 symptom score achieving clinically significant deterioration on QOL. Participants were considered as deteriorated for a given symptom if the change in score from Baseline was 10 points or higher at any time point after Baseline. The data presented is based on the data cut-off date of 21 January 2014 while the study is still ongoing.
Time Frame: as for outcome 9
Population: The analysis was performed using the Intent-to-Treat Population, defined as all randomized subjects.
Measure: Number; unit: Percentage of participants
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Number analyzed (Participants) | 89 | 46
Percentage of participants
  Alopecia (Hair Loss) (N= 80, 39) | 16.3 | 15.4
  Dysphagia (Trouble Swallowing) (N= 80, 39) | 43.8 | 23.1
  Haemoptysis (Coughing Up Blood) (N=80, 39) | 15 | 10.3
  How Much Cough (N=80, 39) | 33.8 | 28.2
  Medicine For Pain (N=43, 21) | 41.9 | 28.6
  Pain In Arm Or Shoulder (N=80, 39) | 55 | 43.6
  Pain In Chest (N=80, 39) | 37.5 | 28.2
  Pain In Other Parts Of Body (N=79, 39) | 51.9 | 38.5
  Peripheral Neuropathy-Tingling Hands/Feet(N=80,39) | 36.3 | 41
  Short Of Breath When Climbed Stairs (N=80, 39) | 45 | 46.2
  Short Of Breath When Rested (N=80, 39) | 36.3 | 41
  Short Of Breath When Walked (N=80, 39) | 45 | 51.3
  Sore Mouth Or Tongue (N=80, 39) | 60 | 5.1

11. Secondary Outcome: Pharmacokinetic (PK) Profile of Lenvatinib in Subjects With Non Small Cell Lung Cancer (NSCLC)
Description: Blood samples were collected for lenvatinib PK analysis. Lenvatinib concentrations from sparse PK sampling were measured. The data is presented as mean nanograms per milliliter +/- Standard deviation of lenvatinib serum concentration.
Time Frame: Cycle 1/Day 1 (between 0.5 and 4 hours postdose and 6 and 10 hours postdose), Cycle 1/Day 15 (predose, between 0.5 and 4 hours postdose, and 6 and 10 hours postdose), and Day 1 of Cycles 2 though 4 (predose and between 2 and 12 hours postdose)
Population: The analysis was performed using the pharmacokinetic (PK) analysis set defined as all subjects who received at least one dose of study drug and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Lenvatinib
Number analyzed (Participants) | 67
nanograms per milliliter
  Cycle 1 Day 1 (0.5 to 4 hours postdose); N=47 | 93.4 (125.66)
  Cycle 1 Day 1 (6 to 10 hours postdose); N=46 | 229.0 (114.06)
  Cycle 1 Day 15 (Pre-dose); N=43 | 77.8 (84.73)
  Cycle 1 Day 15 (0.5 to 4 hours postdose); N=44 | 134.3 (119.44)
  Cycle 1 Day 15 (6 to 10 hours postdose); N=39 | 230.7 (106.29)
  Cycle 2 Day 1 (Pre-dose); N=42 | 68.6 (73.53)
  Cycle 2 Day 1 (2 to 12 hours postdose); N=41 | 260.4 (176.26)
  Cycle 3 Day 1 (Pre-dose); N=34 | 53.5 (49.20)
  Cycle 3 Day 1 (2 to 12 hours postdose); N=31 | 255.3 (173.79)
  Cycle 4 Day 1 (Pre-dose); N=29 | 46.2 (34.94)
  Cycle 4 Day 1 (2 to 12 hours postdose); N=27 | 217.7 (167.70)

ADVERSE EVENTS:
Time Frame: For each participant, from the first dose till 30 days after the last dose or up to approximately 2 years (data cut-off date of 21 January 2014)
Description: Treatment emergent adverse events (TEAEs), defined as an AE (serious/non-serious) that started/increased in severity on/after the first dose of study medication up to 30 days after the final dose of study medication are presented in this section.
Arm/Group | Lenvatinib | Lenvatinib Matched Placebo
Serious Adverse Events (participants affected / at risk) | 46/89 | 21/46
Other Adverse Events (participants affected / at risk) | 83/89 | 42/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib (N=89) | Lenvatinib Matched Placebo (N=46)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 1 | 0
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 4 | 3
CHEST PAIN (General disorders) | 3 | 1
ASTHENIA (General disorders) | 2 | 0
PERFORMANCE STATUS DECREASED (General disorders) | 2 | 0
FATIGUE (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 7 | 3
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 1
SEPSIS (Infections and infestations) | 2 | 0
BRONCHITIS (Infections and infestations) | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0
INFECTION (Infections and infestations) | 1 | 0
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
CACHEXIA (Metabolism and nutrition disorders) | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 0
QUADRIPARESIS (Nervous system disorders) | 1 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
HALLUCINATION (Psychiatric disorders) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 3 | 1
BRONCHIAL POLYP (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 | 0
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib (N=89) | Lenvatinib Matched Placebo (N=46)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 | 0
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 15 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 | 1
CONSTIPATION (Gastrointestinal disorders) | 17 | 8
DIARRHOEA (Gastrointestinal disorders) | 27 | 3
DRY MOUTH (Gastrointestinal disorders) | 7 | 2
DYSPEPSIA (Gastrointestinal disorders) | 13 | 1
NAUSEA (Gastrointestinal disorders) | 26 | 6
STOMATITIS (Gastrointestinal disorders) | 27 | 4
VOMITING (Gastrointestinal disorders) | 23 | 3
ASTHENIA (General disorders) | 16 | 1
CHEST PAIN (General disorders) | 8 | 6
FATIGUE (General disorders) | 24 | 8
MALAISE (General disorders) | 5 | 0
MUCOSAL INFLAMMATION (General disorders) | 5 | 0
OEDEMA PERIPHERAL (General disorders) | 9 | 2
PAIN (General disorders) | 1 | 3
PYREXIA (General disorders) | 10 | 4
PLATELET COUNT DECREASED (Investigations) | 7 | 0
WEIGHT DECREASED (Investigations) | 13 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 31 | 11
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 17 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 | 3
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 5 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 8 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 10 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 1
HEADACHE (Nervous system disorders) | 17 | 6
LETHARGY (Nervous system disorders) | 7 | 2
ANXIETY (Psychiatric disorders) | 4 | 3
INSOMNIA (Psychiatric disorders) | 7 | 3
PROTEINURIA (Renal and urinary disorders) | 33 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 | 10
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 19 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 16 | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 7 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 4
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 9 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 14 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 9 | 1
RASH (Skin and subcutaneous tissue disorders) | 5 | 2
HYPERTENSION (Vascular disorders) | 40 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other